CLINICAL TRIAL: NCT02981485
Title: Fat Grafting Used for the Treatment of Breast Cancer Related Lymphedema in China
Acronym: FGTBRCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Minqiang Xin, Principal Investigator, Peking Union Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZ2015009
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer Lymphedema
Keywords: Fat Grafting, Breast Cancer Lymphedema
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental): Treatment of breast cancer related lymphedema by fat grafting
  Interventions: Device: Fat Grafting

INTERVENTIONS:
Device: Fat Grafting — Treatment of breast cancer related lymphedema by fat grafting

SUMMARY:
Breast cancer related lymphedema (BRCL) is a common complication following breast cancer treatment. The incidence of BRCL ranges from 6-50%, depending on the surgical procedure in the axilla and the type of the radiation therapy. BRCL can causes cosmetic deformities, impaired physical mobility, mental discomfort, reduced quality of life and erysipelas. Therapy of BRCL is divided into conservative and operative methods. However, all the above method has some shortcomings. It is urgent to investigate new approaches to treat BRCL. In this study, fat grafting is to be used for the treatment of BRCL, and the efficacy and safety of this method will be also assessed.

ELIGIBILITY:
Inclusion Criteria:

Breast cancer diagnosis regardless of the date of operation and identified unilateral arm lymphedema Stage Ⅱ of lymphedema according to the standard of International Society of Lymphology The patient is able to read, understand, and complete questionnaires. Completed radiotherapy and/or chemotherapy at least 2 months prior to inclusion The patient understands the nature and purpose of this study and the study procedures and has signed informed consent.

Exclusion Criteria:

Relapse of breast cancer Untreated infection Untreated heart failure Untreated renal failure Untreated deep venous thrombosis in the arm Iodine allergy Pregnancy Psychiatric disorders

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Change in arm volume | Baseline, 3 months, 6months and 12 months
  All the patients who received treatment are scanned by 3 dimensional camera, then the volume measurement of the affected and normal arm is managed by software

SECONDARY OUTCOMES:
Change in tissue edema | Baseline, 3 months, 6months and 12 months
  The affected and normal arms of the patients who received treatment are assessed by multi-frequency bioelectrical impedance analysis
The function of the lymphatic vessel | Baseline, 3 months, 6months and 12 months
  The affected arms of the patients who received treatment was assessed by indocyanine green lymphography
Side effects of treatment | Baseline, 3 months, 6months and 12 months
  Any side effects of experimental treatment. The patients who received treatment are asked at each visit
Change in quality of life | Baseline and 12 months
  The patients who received treatment are asked to fill in a questionnaire (EQ-5D- 5 L-questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Jie Luan, MD, Study Director — Plastic Surgery Hospital of Chinese Academy of Medical Sciences, Peking Union Medical College
Locations (1):
- Plastic Surgery Hospital of Chinese Academy of Medical Sciences, Peking Union Medical College, Shijingshan, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No